CLINICAL TRIAL: NCT06921759
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Lebrikizumab in Adult and Adolescent Participants With Moderate-to-Severe Atopic Hand and Foot Dermatitis
Brief Title: A Study to Investigate the Efficacy and Safety of Lebrikizumab in Participants With Moderate-to-Severe Atopic Hand and Foot Dermatitis
Acronym: ADtouch
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27349; J2T-MC-KGCD (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-04; First posted 2025-04-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atopic Hand and Foot Dermatitis
MeSH Terms: interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lebrikizumab (Experimental): Lebrikizumab administered subcutaneously (SC).
  Interventions: Drug: Lebrikizumab
- Placebo (Placebo Comparator): Placebo Administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150
  Arms: Lebrikizumab
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the efficacy of lebrikizumab versus placebo on skin lesions in adults and adolescent participants with atopic hand and foot dermatitis.

This study lasts up to 32 weeks, including a 6-week screening period, a 16-week treatment period, and a safety follow-up visit 12 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Have an unequivocal diagnosis of chronic atopic hand and/or foot dermatitis at least 1 year prior to screening, regardless of the extent and severity of concomitant atopic dermatitis (AD) on other areas of the body. AD must be present in at least 2 of the 4 mentioned anatomical areas: left hand, right hand, left foot, or right foot at screening and baseline.
* Have a Hand Foot - Investigator Global Assessment (HF-IGA) score of 3 or 4 at the screening and baseline visits.
* Have a baseline hand and foot peak pruritus (numeric rating scale) NRS score ≥4.
* Have a documented history by the investigator of inadequate response to topical medication(s) (topical corticosteroids (TCIs/TCS), topical PDE-4 inhibitors, or topical janus kinase (JAK) inhibitors) in the treatment of atopic hand foot dermatitis (AHFD) within 6 months of screening, or use of topical medications is medically inadvisable (due to intolerance to treatment, hypersensitivity reactions, significant skin atrophy of hand and feet, and systemic effects, as assessed by the investigator or by the treating physician of the participant).
* For adolescent participants, body weight ≥40 kilograms (kg) at baseline.

Exclusion Criteria:

* Have a positive patch test reaction to 1 or more allergens (a score of 1+ or above according to the International Contact Dermatitis Research Group grading scale) before baseline AND which are deemed to be clinically relevant in the view of the investigator as the current cause of the hand and foot dermatitis.
* Have a documented diagnosis of allergic contact dermatitis (ACD) of hands and/or feet, and have a positive patch test reaction at screening, regardless of whether the history of current skin exposure to products containing this allergen (current relevance) is present.
* Have a documented or strong clinical suspicion of the diagnosis of protein contact dermatitis of hands and/or feet. These are the participants with occupational or nonoccupational contact with proteins such as food, latex, and so on, who have positive prick test results and present with lesions of contact urticaria or dermatitis on hands and feet.
* Have a documented exposure to irritants in the occupational or non-occupational (household/recreational) setting that is believed to be a predominant cause of the current hand and foot dermatitis as per the judgment of the investigator.
* Presence of skin comorbidities on hand and/or foot that may interfere with study assessments, such as (but not limited to) palmoplantar psoriasis, palmoplantar keratoderma, impetiginized eczema, lichen planus, pityriasis rubra pilaris, herpes simplex, erythema multiforme, tinea, or scabies.
* Have skin comorbidities that may interfere with study assessments.
* Treatment with topical medications on the hands and feet within 2 weeks before the baseline visit (except for the use of the participant's own emollients).
* Prior treatment with interleukin-13 (IL-13) inhibitors such as lebrikizumab or tralokinumab.
* Have received any live attenuated vaccine within less than 4 weeks of the baseline visit or intend to receive a live attenuated vaccine during the study, or within 4 weeks after receiving the last dose of study intervention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Hand and Foot Investigator Global Assessment (HF-IGA) Score of 0 or 1 with ≥2-point Improvement from Baseline | Week 16
  The HF-IGA is an assessment scale used to determine the severity of hand and foot atopic dermatitis (AD) and clinical response to treatment on a 5-point scale, 0 (clear) to 4 (severe). Higher scores indicate more disease severity.

SECONDARY OUTCOMES:
Percentage of Participants with a HF-Peak Pruritus Numeric Rating Score (NRS) of ≥4 points at Baseline Who Achieve a ≥4-point Reduction (Improvement) from Baseline | Week 16
  The HF-peak pruritus NRS scale is an assessment tool used daily by the participants to rate their worst hand and feet itch intensity on a scale ranging from 0 (no itch) to 10 (worst imaginable itch).
Percentage of Participants with a HF-Peak Pruritus Numeric Rating Score (NRS) of ≥4 points at Baseline Who Achieve a ≥4-point Reduction (Improvement) from Baseline | Week 2
  The HF-peak pruritus NRS scale is an assessment tool used daily by the participants to rate their worst hand and feet itch intensity on a scale ranging from 0 (no itch) to 10 (worst imaginable itch).
Percentage of Participants with HF-Peak Pruritus NRS of ≥4 points at Baseline Who Achieve a ≥4-point Reduction (Improvement) from Baseline | Baseline, Week 4
  The HF-peak pruritus NRS scale is an assessment tool used daily by the participants to rate their worst hand and feet itch intensity on a scale ranging from 0 (no itch) to 10 (worst imaginable itch).
Percentage of Participants with a HF-Peak Pain NRS of ≥4 points at Baseline Who Achieve a ≥4-point Reduction (Improvement) from Baseline | Week 16
  The HF-peak pain NRS Scale is an assessment tool used daily by the participants to report the intensity of pain. Participants select the number between 0 and 10 that best fits their worst pain intensity over the past 24 hours (0 = no pain and 10 = the worst pain possible).
Percentage of Participants Achieving a Hand and Foot Investigator Global Assessment (HF-IGA) Score of 0 or 1 with ≥2-point Improvement from Baseline | Week 4
  The HF-IGA is an assessment scale used to determine the severity of hand and foot atopic dermatitis (AD) and clinical response to treatment on a 5-point scale, 0 (clear) to 4 (severe). Higher scores indicate more disease severity.
Percentage of Participants Achieving a Hand and Foot Investigator Global Assessment (HF-IGA) Score of 0 or 1 with ≥2-point Improvement from Baseline | Week 8
  The HF-IGA is an assessment scale used to determine the severity of hand and foot atopic dermatitis (AD) and clinical response to treatment on a 5-point scale, 0 (clear) to 4 (severe). Higher scores indicate more disease severity.
Percentage of Participants Who Are "Satisfied" or "Very Satisfied" on Atopic Hand Dermatitis Clearance Satisfaction (AHDCS) | Week 16
  This single-item question assesses participants' satisfaction with hand clearance at the current time. The response options are reported as the percentage of participants who selected 1 of the following: Very Satisfied, Satisfied, Neither Satisfied nor Dissatisfied, Dissatisfied, or Very Dissatisfied.
Percent Change from Baseline in Hand and Foot Peak Pain NRS | Baseline, Week 16
  The HF-peak pain NRS Scale is an assessment tool used daily by the participants to report the intensity of pain. Participants select the number between 0 and 10 that best fits their worst pain intensity over the past 24 hours (0 = no pain and 10 = the worst pain possible).
Percent Change from Baseline in Modified Total Lesion Symptom Scale (mTLSS) for Hand and Foot Lesions | Baseline, Week 16
  The mTLSS is an investigator-reported scale that combines the evaluation of lesion severity of hand eczema (HE) (erythema, edema, desquamation, fissures, hyperkeratosis or lichenification, and vesicles) with the intensity of pruritus or pain to assess the severity of symptoms. This composite score assigns 0 (mild) to 3 (severe) to each component, giving a maximum disease severity of 21. A separate score is assigned for hands and feet.
Percentage of Participants with Hand Dermatitis Achieving HECSI-90 Score | Week 16
  The HECSI scoring system incorporates both the extent and the intensity of the disease. The total sum called the HECSI score will be calculated, varying from 0 to a maximum severity score of 360 points.
Percent Change from Baseline in Hand Eczema Severity Index (HECSI) Score for Participants with Hand Dermatitis | Baseline, Week 16
  The HECSI scoring system incorporates both the extent and the intensity of the disease. The total sum called the HECSI score will be calculated, varying from 0 to a maximum severity score of 360 points.
Percentage of Participants with Hand Dermatitis Achieving HECSI-50 Score | Week 16
  The HECSI scoring system incorporates both the extent and the intensity of the disease. The total sum called the HECSI score will be calculated, varying from 0 to a maximum severity score of 360 points.
Percentage of Participants with Hand Dermatitis Achieving HECSI-75 Score | Week 16
  The HECSI scoring system incorporates both the extent and the intensity of the disease. The total sum called the HECSI score will be calculated, varying from 0 to a maximum severity score of 360 points.
Change from Baseline in Quality of Life in Hand Eczema Questionnaire (QOLHEQ) for Participants with Hand Dermatitis | Baseline, Week 16
  The QOLHEQ consists of 30 items that can be summarized according to 4 domains of HRQoL: impairments over the last 7 days because of (1) symptoms, (2) emotions, (3) limitations in functioning, or (4) treatment and prevention. The total QOLHEQ score ranges between 0 and 117, with higher scores indicative of a poor HE-specific HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (79):
- United States (14):
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Encore Medical Research, Hollywood, Florida
  - Research Associates of South Florida - Miami - Southwest 8th Street, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - DeNova Research, Chicago, Illinois
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Revival Research Institute, LLC, Troy, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Care Access - Hoboken, Hoboken, New Jersey
  - Optima Research - Boardman, Boardman, Ohio
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Complete Dermatology, Sugar Land, Texas
- Argentina (11):
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - CIPREC, Buenos Aires
  - Instituto de Neumonologia Y Dermatologia, Buenos Aires
  - Psoriahue, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Parra Dermatología, Mendoza
  - Fundacion Estudios Clinicos, Rosario
  - INECO Neurociencias Oroño, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Centro de Investigaciones San Miguel, San Miguel
- Australia (8):
  - The Skin Centre, Benowa
  - Skin Health Institute Inc., Carlton
  - Cornerstone Dermatology, Coorparoo
  - Fremantle Dermatology, Fremantle
  - St George Dermatology & Skin Cancer Centre, Kogarah
  - Institute for Skin, Health and Immunity, Mitcham
  - Paratus Clinical Research Woden, Phillip
  - Veracity Clinical Research, Woolloongabba
- Canada (10):
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie
  - INTERMED Groupe Sante, Chicoutimi
  - Interior Dermatology Centre - Probity - PPDS, Kelowna
  - DermEffects, London
  - Centre de Recherche Saint-Louis, Montreal
  - Centre de Recherche Saint-Louis, Québec
  - CaRe Clinic, Red Deer
  - Private Practice - Dr. Rachel Asiniwasis, Regina
  - FACET Dermatology, Toronto
  - Wiseman Dermatology Research Inc., Winnipeg
- Japan (8):
  - Kosugi Dermatology Clinic, Kawasaki-shi
  - Maruyama Dermatology Clinic, Kōtoku
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Tanpopo Skin Clinic, Ōta-ku
  - Pansy Skin Clinic, Saitama
  - Dermatology and Ophthalmology Kume Clinic, Sakai
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Tachikawa Dermatology Clinic, Tachikawa
- Mexico (8):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Ciudad de México
  - Grupo Clínico CATEI S.C., Guadalajara
  - RM Pharma Specialists, Mexico City
  - Kohler & Milstein Research S.A. De C.V., Mérida
  - Eukarya Pharmasite S.C., Monterrey
  - Arké SMO S.A de C.V, Veracruz
  - Instituto Dermatologico de Jalisco, Zapopan
- South Korea (12):
  - Korea University Ansan Hospital, Ansan-si
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Bupyeong-gu
  - Pusan National University Yangsan Hospital, Busan
  - Chosun University Hospital, Gwangju
  - Kyungpook National University Hospital, Junggu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (8):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - New Taipei Municipal TuCheng Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
  - National Taiwan University Hospital - Hsinchu branch, Zhubei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Lilly Trials — http://trials.lilly.com/en-US/trial/591896